CLINICAL TRIAL: NCT03435367
Title: Immersive Virtual Reality to Reduce Procedural Pain During IV Insertion in Children in the Emergency Department: A Feasibility Pilot Study
Brief Title: Immersive Virtual Reality to Reduce Procedural Pain During IV Insertion in Children in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000058799
Record Dates: First submitted 2018-01-19; First posted 2018-02-19 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: IV Insertion in the Emergency Department

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (VR) (Experimental): The patient will be allowed to 'try-out' the VR system (including all auditory and visual features) for ~5 minutes prior to the start of the procedure. In addition to usual care, consisting of child-life presence and topical analgesics if ordered by the treating medical team, children in the experimental condition will wear the VR HMD plus headphones and hold the VR controller.
  Interventions: Device: Virtual Reality Program
- Control Group (Standard Care - Video) (Active Comparator): The patient will be allowed to watch an age-appropriate video on a tablet device. The patient will be offered to wear the same headphones as in the experimental condition. The patient will have the tablet and headphones for ~5 minutes prior to the start of the procedure. In addition, the patient will receive standard care consisting of a child life specialist and topical analgesics (if ordered by the treating medical team).
  Interventions: Device: iPad Tablet

INTERVENTIONS:
Device: Virtual Reality Program — VR with head mounted display (HMD) and headphones.
  Arms: Intervention Group (VR)
Device: iPad Tablet — iPad with headphones
  Arms: Control Group (Standard Care - Video)

SUMMARY:
Venipuncture and intravenous (IV) access continue to be the most common causes of pain and distress among children in the pediatric emergency department. Virtual reality has been successful for reducing pain and fear in many clinical scenarios, including port access in oncology patients, anxiety disorders, phobias, burn and wound care and others. There is only one previous study examining virtual reality distraction to reduce procedural pain during IV insertion in pediatric patients and no previous studies examining this in the emergency department setting. In this study, the investigators will compare immersive virtual reality (an interactive underwater environment) to the current standard (tablet device/iPad playing a movie) for distraction to reduce procedural pain during IV insertion. The investigators hypothesize that the immersive quality of the virtual reality will reduce patient's pain scores, fear scores and tachycardia during and after the procedure, and have minimal effect on departmental flow and nursing satisfaction. If this feasibility pilot study yields positive results, the investigators plan to expand to a larger randomized control trial.

DETAILED DESCRIPTION:
This study is a pilot randomized control trial that aims to (a) to determine the differences in self-reported and proxy-reported pain and fear during IV insertion between the interactive VR intervention and control group, and (b) to assess the feasibility (safety, acceptability) of the VR intervention to children/families and the healthcare team in the pediatric emergency department. The study will consist of two study arms, where both study arms will be screened and recruited using the same procedure. Participants will be randomized into either (1) Control group: child life specialist plays an age-appropriate video on a tablet device, or (2) Intervention (VR Distraction): child life specialist facilitates immersive VR experience. Both the intervention and control groups will receive standard medical care (e.g., topical anesthetics). A convenience sample of 80 children and adolescents with cancer (40 participants per treatment arm; 20 boys and 20 girls per treatment arm) will be recruited. In addition to usual care, children in the experimental condition will wear the VR headset plus headphones. In the control condition, children will watch a video (i.e., an age-appropriate video selected by an emergency department affiliated child life specialist) on an iPad, while wearing the same headphones as in the experimental condition. Implementation outcomes include accrual and retention rates, acceptability and technical difficulties. Effectiveness outcomes include child pain, distress, and fear, as well as parent distress.

ELIGIBILITY:
Inclusion criteria will be:

1. aged 8-17 years
2. able to speak and understand English
3. parent/guardian present
4. medically stable (CTAS 2, 3, 4 or 5; IV insertion +/-20 minutes will not impact the safety of the patient according to treating medical team)
5. requires IV insertion

Exclusion criteria will be:

1. visual, auditory or cognitive impairments precluding interaction with the VR intervention or reporting pain and fear
2. psychiatric conditions that could be exacerbated by the VR environment (i.e. hallucinations)
3. skin, face or ear infections or injuries, which could contaminate the intervention equipment
4. medically unstable (CTAS 1; patient requires immediate IV insertion)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline, 30 minutes after baseline
  Using an 11 point Numerical Rating Scale (NRS) (0 being no distress at all and 10 being the most distress you can imagine this child or you having) children will self-report their pain and parents, nurses and the researcher will report children's pain BOTH prior to and following the procedure.
Change in Child Distress | Baseline, 30 minutes after baseline
  Using an 11 point Numerical Rating Scale (NRS) (0 being no distress at all and 10 being the most distress you can imagine this child or you having) children will self-report their distress and parents, nurses and the researcher will report children's distress BOTH prior to and following the procedure
Change in Child Fear | Baseline, 30 minutes after baseline
  Children will report fear BOTH prior to and following the procedure using the Child Fear Scale (CFS) which is a 5-face visual scale that measures fear intensity and is validated in children as young as 5 years. It consists of a 1-question scale rating fear from 0 - 4, based on the faces provided. A higher number represents higher fear intensity.
Child Pain Catastrophizing | Baseline
  Children will report baseline tendencies to catastrophize about pain using the Pain Catastrophizing Scale - Child (PCS-C). This is a self-report measure of children's tendency to catastrophize about pain validated in children 8-18 years of age. 6-items responded to on an 11-point scale from 0 ("not at all") to 10 ("a lot"), with a higher number representing higher pain catastrophizing.
Parent Pain Catastrophizing | Baseline
  Parents will report baseline tendencies to catastrophize about their child's pain using the Pain Catastrophizing Scale - Parent (PCS-P), which is a self-report measure of parents' tendency to catastrophize about their child's pain validated in parents of children 8-18 years of age. 6-items responded to on an 11-point scale from 0 ("not at all") to 10 ("a lot"), with a higher number representing higher parental pain catastrophizing of their child's pain.
Parent Distress | 30 minutes after baseline measures are completed
  Parents will report on their own level of distress following the child's procedure using the Parent Distress Questionnaire. This measure consists of 4-items responded to on an 11-point numeric rating scale from 0 ("not at all") to 10 ("extremely"). A higher number value represents higher distress levels.
Child Presence Measure | 30 minutes after baseline measures are completed
  This child self-report measure assesses effectiveness of the immersive aspect of the VR toolkit/iPad using 12 questions, a choice of three answers ("no", "a little", and "a lot").

SECONDARY OUTCOMES:
Recruitment log | through study completion, an average of 1 year
  Using an investigator-generated recruitment log, accrual rates will be measured by counting the number eligible children per recruitment day, participants enrolled, reasons for ineligibility, reasons for non-participation and reasons for study attrition.
Acceptability | 30 minutes after baseline measures are completed
  Measured using the VR Distraction Satisfaction Questionnaire completed by children, parents and nurses and will collect data on acceptability, perceived utility of pain reducing procedures, and recommendations for changes related to the needle insertion experience.
Outcome measure feasibility | through study completion, an average of 1 year
  Will be measured as the percentage of completed outcome measures at baseline and study completion and will be recorded on the VR Distraction Activity Log.
Technical Difficulties Log | through study completion, an average of 1 year
  Using an investigator-generated technical difficulties log, researchers will record data related to technical difficulties associated with the VR intervention, observed difficulties in implementing the trial protocol in the clinic and time to complete IV needle insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada